CLINICAL TRIAL: NCT01176097
Title: A Randomized, Single-Blind, Placebo-Controlled, Single-Center, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and the Effect of Fasting After Single Ascending Oral Doses of AZD5658 in Type 2 Diabetes Mellitus Patients
Brief Title: To Assess Safety, Tolerability, Pharmacokinetics/Pharmacodynamics and the Effect of Fasting After Single Oral Doses of AZD5658 in Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: D2920C00001
Record Dates: First submitted 2010-07-19; First posted 2010-08-05 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes
Keywords: First in man study evaluating AZD5658 in Type 2 Diabetics.; Effect of fasting; Safety; Tolerability
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 6 - 8 cohorts (Experimental): 6 patients in each cohort will receive AZD5658
  Interventions: Drug: AZD5658; Drug: Placebo
- 6 - 8 cohorts (Placebo Comparator): 2 patients in each cohort will receive placebo
  Interventions: Drug: AZD5658; Drug: Placebo

INTERVENTIONS:
Drug: AZD5658 — oral suspension, escalating single doses
Drug: Placebo — oral suspension,single doses

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of AZD5658 following ascending single oral doses in Type 2 Diabetics. It will also estimate the maximum tolerated dose.

DETAILED DESCRIPTION:
This is a randomized, single-blind, placebo-controlled, single-center, phase 1 study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and the effect of fasting after single ascending oral doses of AZD5658 in type 2 diabetes mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be of non-childbearing potential.
* Body mass index between greater than or equal to 19 and less than or equal to 40 kg/m2
* Patients with confirmed Type 2 Diabetes diagnosis for at least 1 year and treated with Metformin

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma within 2 weeks before the first administration of the IP
* Participation in another clinical study during the last 30 days prior to enrollment
* Significant cardiovascular event within the last 6 months prior to enrollment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of AZD5658 following oral administration of single ascending doses and to estimate the maximum tolerated dose (MTD). | AEs-, blood pressure and pulse during study days. Safety labs - day -1 to day 4; ECG - days 1, 2 and 3

SECONDARY OUTCOMES:
To investigate the pharmacokinetics of AZD5658 after single ascending oral doses in type 2 diabetes mellitus patients. | Venous blood samples for the determination of concentrations of AZD5658 in plasma will be taken predose and at various times up to 72 hours postdose
Pharmacodynamics (plasma glucose and serum insulin) | Plasma glucose and serum insulin determined on Day -1 through Day 4
Effect of fasting on the pharmacokinetics and explore the pharmacodynamics of AZD5658.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Wahlander, Study Director — AstraZeneca R&DPepparedsleden 1431 83 M�lnda; Mirjana Kujacic, Study Chair — AstraZeneca R&DPepparedsleden 1431 83 M�lndal; Linda Morrow, Principal Investigator — Profil Institute for Clinical Research, Inc.855 Third Avenue, Suite 4400Chula Vista, CA 91911
Locations (1):
- Research Site, Chula Vista, California, United States